CLINICAL TRIAL: NCT03145701
Title: Predicting Cerebral Aneurysm Recurrence Using Doppler Guidewire Measurements
Brief Title: Doppler Flow Wires in Cerebral Angiography
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Louis Kim, Professor, Neurological Surgery, University of Washington
Other Study IDs: STUDY00002026
Record Dates: First submitted 2017-04-06; First posted 2017-05-09 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Aneurysm; Cerebral Aneurysm
MeSH Terms: conditions — Aneurysm; Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to use a wire with a Doppler tip to measure blood flow in vessels in the brain and determine hemodynamic factors associated with treatment success or failure. Many neurological diseases cause abnormal blood flow in the brain in specific vessels. The special wire used in this study is place into brain blood vessels during standard of care procedure to treat such diseases, and blood flow parameters (such as velocity and pressure) are measured to gain better understanding of these neurological diseases.

DETAILED DESCRIPTION:
Current treatments of cerebral aneurysms are imperfect, and aneurysmal hemodynamics is an important factor in treatment failure. The identification of hemodynamic factors that influence treatment success could predict outcome. Published studies show that the hemodynamic environment of aneurysms changes after treatment, and there is limited retrospective evidence that the degree of change affects treatment success. However, previous hemodynamic calculations did not have access to patient-specific measurements of blood flow, which substantially reduced their accuracy. In addition, no prospective studies of the predictive value of post-treatment aneurysm hemodynamics have been done.

Methods: Prospectively test new aneurysm patients for hemodynamic predictors of treatment outcome based upon the hypothesis long-term aneurysm treatment outcome can be prospectively predicted by measuring the immediate hemodynamic effects of aneurysm treatment with novel patient-specific modeling techniques. Task 1: In a new cohort of patients undergoing aneurysm treatment, the investigators will again use Doppler guidewire measurements to create patient-specific hemodynamic models of treatment effects. By prospectively applying the knowledge of crucial hemodynamic changes the investigators will use immediate post-treatment hemodynamics to predict long-term treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an unruptured intracranial aneurysm ≥ 5mm in size undergoes endovascular treatment and subsequent angiographic follow-up

Exclusion Criteria:

-previously enrolled in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be eligible for this aim if they were not previously enrolled in the study, as this phase seeks to prospectively apply the tests generated by the previous retrospective cohort. Selection criteria will be similar in which a patient with an unruptured intracranial aneurysm ≥ 5mm in size undergoes endovascular treatment and subsequent angiographic follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Treatment Prediction | May 2017- July 2019
  The results of this prospective aim have the potential to substantially influence aneurysm management by predicting long-term outcome at the time of initial treatment. The investigators will determine how well the prospective test predicts long-term treatment success as applied at the time of treatment, using computational fluid dynamics modeling of hemodynamic factors with the incorporation of patient-specific measurements obtained by the Doppler guidewire

CONTACTS AND LOCATIONS:
Overall Officials: Louis J Kim, MD, Principal Investigator — University of Washington Department of Neurological Surgery
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No